CLINICAL TRIAL: NCT04043780
Title: Clinical Validation of a Decompression Prototype Splint for Patients With Carpal Tunel Syndrome: a Multicentric Randomized Controlled Trial
Brief Title: Clinical Validation of a Decompression Prototype Splint for Patients With Carpal Tunel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: Salud Aragon (Unknown); Universitat de Catalunya (Unknown); Institut Català de la Salut (Other)
Responsible Party: Principal Investigator, Elena Estebanez de Miguel, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI19/334
Record Dates: First submitted 2019-07-30; First posted 2019-08-02 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decompression prototype splint (Experimental): The patients of this group will wear the decompression prototype splint.
  Interventions: Device: Decompression prototype splint for carpal tunnel syndrome
- standard splint (Active Comparator): The patients of this group will wear a standard splint.
  Interventions: Device: Standard splint for carpal tunnel syndrome

INTERVENTIONS:
Device: Decompression prototype splint for carpal tunnel syndrome — This group will wear during 6 weeks a decompression prototype splint. They we be informed to wear it as long as possible during the 6 weeks.
  Arms: Decompression prototype splint
Device: Standard splint for carpal tunnel syndrome — This group will wear during 6 weeks a standard splint. They we be informed to wear it as long as possible during the 6 weeks.
  Arms: standard splint

SUMMARY:
A multicentric randomized controlled trial has been designed to study the effects of a decompression prototype splint on symptoms, functional capacity and nerve conduction studies in patients with carpal tunnel syndrome.

DETAILED DESCRIPTION:
A decompression prototype splint was designed to simulate an manual mobilization that is able to increase the CSA of the carpal tunnel and the median nerve in cadavers. These changes are important because they may relate to the decrease in CTS symptoms.

Patients with mild or moderate carpal tunnel syndrome will be selected for the trial. They will be randomized in 2 groups. One group will wear an standard splint for carpal tunnel syndrome and the other the decompression prototype splint.

ELIGIBILITY:
Inclusion Criteria:

* Be medically diagnosed with carpal tunnel syndrome after electrophysiological tests and present mild to moderate involvement. This test is performed according to the standards established by the "American Academy of Physical Medicine and Rehabilitation"
* Ability to understand and communicate their symptoms and to complete the questionnaires.

Exclusion Criteria:

* Previous surgery in the carpal tunnel in the same limb Other pathologies that may be associated with carpal tunnel syndrome: traumas, pathologies or disorders of the upper limb or cervical spine (cervical radiculopathy, cervical sprain, etc.) or prior cervical surgery
* Concurrent comorbidities that may be the cause and interfere with the treatment of the carpal tunnel syndrome: diabetes mellitus, hypothyroidism, rheumatoid arthritis, fibromyalgia, reflex sympathetic dysfunction, obesity, renal disease, alcoholism, significant vitamin deficiency and associated viral or bacterial processes
* Pregnancy
* Oral drugs, physiotherapy treatment , treatment with splints or infiltrations for carpal tunnel syndrome prior or during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Intensity of symptoms at baseline | Baseline
  Intensity of the symptoms (pain, paraesthesia...) will be assess with a visual analogic scale (VAS). A VAS is usually a 100-mm long horizontal line with verbal descriptors (word anchors) at each end to express the extremes of the feeling. Patients mark the point on the line that best corresponds to their symptom severity . When reading the VAS, the position of the respondent's cross is generally assigned a score between 0 and 100. The scores can then be simply transferred to a 100-value scale using a millimeter tape measure.
Intensity of the symptoms at 6 weeks | 6 weeks
  Intensity of the symptoms (pain, paraesthesia...) will be assess with a visual analogic scale (VAS). A VAS is usually a 100-mm long horizontal line with verbal descriptors (word anchors) at each end to express the extremes of the feeling. Patients mark the point on the line that best corresponds to their symptom severity . When reading the VAS, the position of the respondent's cross is generally assigned a score between 0 and 100. The scores can then be simply transferred to a 100-value scale using a millimeter tape measure.
Intensity of the symptoms at 4 months | 4 months
  Intensity of the symptoms (pain, paraesthesia...) will be assess with a visual analogic scale (VAS). A VAS is usually a 100-mm long horizontal line with verbal descriptors (word anchors) at each end to express the extremes of the feeling. Patients mark the point on the line that best corresponds to their symptom severity . When reading the VAS, the position of the respondent's cross is generally assigned a score between 0 and 100. The scores can then be simply transferred to a 100-value scale using a millimeter tape measure.
Nerve conduction studies at baseline | Baseline
  The nerve conduction will be assess with electroneurogram.
Nerve conduction studies at 6 weeks | 6 weeks
  The nerve conduction will be assess with electroneurogram.
Self-reported symptom severity and functional status at baseline | Baseline
  This outcome will be assess with The Boston Carpal Tunnel Questionnaire (BCTQ), that is a disease-specific measure of self-reported symptom severity and functional status. The Boston Carpal Tunnel Questionnaire (BCTQ), is a patient-based outcome measure that has been developed specifically for patients with CTS. It has two distinct scales, the Symptom Severity Scale (SSS) which has 11 questions and uses a five-point rating scale and the Functional Status Scale (FSS) containing 8 items which have to be rated for degree of difficulty on a five-point scale. Each scale generates a final score (sum of individual scores divided by number of items) which ranges from 1 to 5, with a higher score indicating greater disability.
Self-reported symptom severity and functional status at 6 weeks | 6 weeks
  This outcome will be assess with The Boston Carpal Tunnel Questionnaire (BCTQ), that is a disease-specific measure of self-reported symptom severity and functional status. The Boston Carpal Tunnel Questionnaire (BCTQ), is a patient-based outcome measure that has been developed specifically for patients with CTS. It has two distinct scales, the Symptom Severity Scale (SSS) which has 11 questions and uses a five-point rating scale and the Functional Status Scale (FSS) containing 8 items which have to be rated for degree of difficulty on a five-point scale. Each scale generates a final score (sum of individual scores divided by number of items) which ranges from 1 to 5, with a higher score indicating greater disability.
Self-reported symptom severity and functional status at 4 months | 4 months
  This outcome will be assess with The Boston Carpal Tunnel Questionnaire (BCTQ), that is a disease-specific measure of self-reported symptom severity and functional status. The Boston Carpal Tunnel Questionnaire (BCTQ), is a patient-based outcome measure that has been developed specifically for patients with CTS. It has two distinct scales, the Symptom Severity Scale (SSS) which has 11 questions and uses a five-point rating scale and the Functional Status Scale (FSS) containing 8 items which have to be rated for degree of difficulty on a five-point scale. Each scale generates a final score (sum of individual scores divided by number of items) which ranges from 1 to 5, with a higher score indicating greater disability.
Global Perceived Effect at 6 weeks | 6 weeks
  Global perceived effect will be assess with the Global Perceived Effect scale. The global perceived effect scale (GPES) is a commonly used method for measuring patients' assessment of their condition. One of the underlying assumptions of the GPE is that it measures a global assessment of change in the patient's chief complaint. Global Perceived Effect Scale (GPES) consists of a scale of five points that varies from less than five points (much worse), zero (no change) and five points (completely recovered). The participants are asked in the following way for all the measures of the overall effect perceived: "Compared with the beginning of the episode, how do you describe your wrist/hand today?". Positive scores represent better recovery and negative scores indicate a worsening of symptoms.
Global Perceived Effect at 4 months | 4 months
  Global perceived effect will be assess with the Global Perceived Effect scale. The global perceived effect scale (GPES) is a commonly used method for measuring patients' assessment of their condition. One of the underlying assumptions of the GPES is that it measures a global assessment of change in the patient's chief complaint. Global Perceived Effect Scale (GPES) consists of a scale of five points that varies from less than five points (much worse), zero (no change) and five points (completely recovered). The participants are asked in the following way for all the measures of the overall effect perceived: "Compared with the beginning of the episode, how do you describe your wrist/hand today?". Positive scores represent better recovery and negative scores indicate a worsening of symptoms.

SECONDARY OUTCOMES:
Adherence to the treatment | 6 weeks
  The participants will fill in a calendar indicating the hours of use

CONTACTS AND LOCATIONS:
Overall Officials: Elena Estébanez-de-Miguel, PhD, Principal Investigator — Universidad de Zaragoza
Locations (1):
- Elena Estébanez de Miguel, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keith MW, Masear V, Chung KC, Maupin K, Andary M, Amadio PC, Watters WC 3rd, Goldberg MJ, Haralson RH 3rd, Turkelson CM, Wies JL, McGowan R. American Academy of Orthopaedic Surgeons Clinical Practice Guideline on diagnosis of carpal tunnel syndrome. J Bone Joint Surg Am. 2009 Oct;91(10):2478-9. doi: 10.2106/JBJS.I.00643. No abstract available. PMID 19797585
- [Background] Werner RA, Andary M. Carpal tunnel syndrome: pathophysiology and clinical neurophysiology. Clin Neurophysiol. 2002 Sep;113(9):1373-81. doi: 10.1016/s1388-2457(02)00169-4. PMID 12169318
- [Background] Atroshi I, Gummesson C, Johnsson R, Ornstein E, Ranstam J, Rosen I. Prevalence of carpal tunnel syndrome in a general population. JAMA. 1999 Jul 14;282(2):153-8. doi: 10.1001/jama.282.2.153. PMID 10411196
- [Background] Buckle PW, Devereux JJ. The nature of work-related neck and upper limb musculoskeletal disorders. Appl Ergon. 2002 May;33(3):207-17. doi: 10.1016/s0003-6870(02)00014-5. PMID 12164505
- [Background] Foley M, Silverstein B, Polissar N. The economic burden of carpal tunnel syndrome: long-term earnings of CTS claimants in Washington State. Am J Ind Med. 2007 Mar;50(3):155-72. doi: 10.1002/ajim.20430. PMID 17216630
- [Background] Foley M, Silverstein B. The long-term burden of work-related carpal tunnel syndrome relative to upper-extremity fractures and dermatitis in Washington State. Am J Ind Med. 2015 Dec;58(12):1255-69. doi: 10.1002/ajim.22540. Epub 2015 Nov 2. PMID 26523842
- [Background] Stapleton MJ. Occupation and carpal tunnel syndrome. ANZ J Surg. 2006 Jun;76(6):494-6. doi: 10.1111/j.1445-2197.2006.03770.x. PMID 16768777
- [Background] Roel-Valdes J, Arizo-Luque V, Ronda-Perez E. [Epidemiology of occupationally-caused carpal tunnel syndrome in the province of Alicante, Spain 1996-2004]. Rev Esp Salud Publica. 2006 Jul-Aug;80(4):395-409. doi: 10.1590/s1135-57272006000400009. Spanish. PMID 16913614
- [Background] Akalin E, El O, Peker O, Senocak O, Tamci S, Gulbahar S, Cakmur R, Oncel S. Treatment of carpal tunnel syndrome with nerve and tendon gliding exercises. Am J Phys Med Rehabil. 2002 Feb;81(2):108-13. doi: 10.1097/00002060-200202000-00006. PMID 11807347
- [Background] Ballestero-Perez R, Plaza-Manzano G, Urraca-Gesto A, Romo-Romo F, Atin-Arratibel MLA, Pecos-Martin D, Gallego-Izquierdo T, Romero-Franco N. Effectiveness of Nerve Gliding Exercises on Carpal Tunnel Syndrome: A Systematic Review. J Manipulative Physiol Ther. 2017 Jan;40(1):50-59. doi: 10.1016/j.jmpt.2016.10.004. Epub 2016 Nov 11. PMID 27842937
- [Background] Baker NA, Moehling KK, Rubinstein EN, Wollstein R, Gustafson NP, Baratz M. The comparative effectiveness of combined lumbrical muscle splints and stretches on symptoms and function in carpal tunnel syndrome. Arch Phys Med Rehabil. 2012 Jan;93(1):1-10. doi: 10.1016/j.apmr.2011.08.013. PMID 22200381
- [Background] Page MJ, Massy-Westropp N, O'Connor D, Pitt V. Splinting for carpal tunnel syndrome. Cochrane Database Syst Rev. 2012 Jul 11;2012(7):CD010003. doi: 10.1002/14651858.CD010003. PMID 22786532
- [Background] Brininger TL, Rogers JC, Holm MB, Baker NA, Li ZM, Goitz RJ. Efficacy of a fabricated customized splint and tendon and nerve gliding exercises for the treatment of carpal tunnel syndrome: a randomized controlled trial. Arch Phys Med Rehabil. 2007 Nov;88(11):1429-35. doi: 10.1016/j.apmr.2007.07.019. PMID 17964883
- [Background] Wang JC, Liao KK, Lin KP, Chou CL, Yang TF, Huang YF, Wang KA, Chiu JW. Efficacy of Combined Ultrasound-Guided Steroid Injection and Splinting in Patients With Carpal Tunnel Syndrome: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 May;98(5):947-956. doi: 10.1016/j.apmr.2017.01.018. Epub 2017 Feb 14. PMID 28209506
- [Background] Manente G, Torrieri F, Di Blasio F, Staniscia T, Romano F, Uncini A. An innovative hand brace for carpal tunnel syndrome: a randomized controlled trial. Muscle Nerve. 2001 Aug;24(8):1020-5. doi: 10.1002/mus.1105. PMID 11439376
- [Background] Li ZM, Gabra JN, Marquardt TL, Kim DH. Narrowing carpal arch width to increase cross-sectional area of carpal tunnel--a cadaveric study. Clin Biomech (Bristol). 2013 Apr;28(4):402-7. doi: 10.1016/j.clinbiomech.2013.02.014. Epub 2013 Apr 9. PMID 23583095
- [Background] Marquardt TL, Gabra JN, Li ZM. Morphological and positional changes of the carpal arch and median nerve during wrist compression. Clin Biomech (Bristol). 2015 Mar;30(3):248-53. doi: 10.1016/j.clinbiomech.2015.01.007. Epub 2015 Jan 31. PMID 25661267
- [Background] Bueno-Gracia E, Ruiz-de-Escudero-Zapico A, Malo-Urries M, Shacklock M, Estebanez-de-Miguel E, Fanlo-Mazas P, Caudevilla-Polo S, Jimenez-Del-Barrio S. Dimensional changes of the carpal tunnel and the median nerve during manual mobilization of the carpal bones. Musculoskelet Sci Pract. 2018 Aug;36:12-16. doi: 10.1016/j.msksp.2018.04.002. Epub 2018 Apr 4. PMID 29635191
- [Background] Bueno-Gracia E, Perez-Bellmunt A, Lopez-de-Celis C, Shacklock M, Salas-Lopez A, Simon M, Alvarez-Diaz P, Tricas-Moreno JM. Dimensional changes of the carpal tunnel and median nerve during manual mobilization of the carpal bones - Anatomical study. Clin Biomech (Bristol). 2018 Nov;59:56-61. doi: 10.1016/j.clinbiomech.2018.09.001. Epub 2018 Sep 3. PMID 30195102
- [Background] Bulut GT, Caglar NS, Aytekin E, Ozgonenel L, Tutun S, Demir SE. Comparison of static wrist splint with static wrist and metacarpophalangeal splint in carpal tunnel syndrome. J Back Musculoskelet Rehabil. 2015;28(4):761-7. doi: 10.3233/BMR-140580. PMID 25547237
- [Background] De Angelis MV, Pierfelice F, Di Giovanni P, Staniscia T, Uncini A. Efficacy of a soft hand brace and a wrist splint for carpal tunnel syndrome: a randomized controlled study. Acta Neurol Scand. 2009 Jan;119(1):68-74. doi: 10.1111/j.1600-0404.2008.01072.x. Epub 2008 Jul 13. PMID 18638040
- [Background] Golriz B, Ahmadi Bani M, Arazpour M, Bahramizadeh M, Curran S, Madani SP, Hutchins SW. Comparison of the efficacy of a neutral wrist splint and a wrist splint incorporating a lumbrical unit for the treatment of patients with carpal tunnel syndrome. Prosthet Orthot Int. 2016 Oct;40(5):617-23. doi: 10.1177/0309364615592695. Epub 2015 Jul 20. PMID 26195619
- [Background] Zinnuroglu M, Baspinar M, Beyazova M. Carpal lock and the volar-supporting orthosis in mild and moderate carpal tunnel syndrome. Am J Phys Med Rehabil. 2010 Sep;89(9):759-64. doi: 10.1097/PHM.0b013e3181e721ed. PMID 20581649
- [Background] Bland JD. A neurophysiological grading scale for carpal tunnel syndrome. Muscle Nerve. 2000 Aug;23(8):1280-3. doi: 10.1002/1097-4598(200008)23:83.0.co;2-y. PMID 10918269
- [Background] Barbosa RI, Fonseca Mde C, Rodrigues EK, Tamanini G, Marcolino AM, Mazzer N, Guirro RR, MacDermid J. Efficacy of low-level laser therapy associated to orthoses for patients with carpal tunnel syndrome: A randomized single-blinded controlled trial. J Back Musculoskelet Rehabil. 2016 Aug 10;29(3):459-66. doi: 10.3233/BMR-150640. PMID 26444330
- [Background] Celik B, Paker N, Celik EC, Bugdayci DS, Ones K, Ince N. The effects of orthotic intervention on nerve conduction and functional outcome in carpal tunnel syndrome: A prospective follow-up study. J Hand Ther. 2015 Jan-Mar;28(1):34-7; quiz 38. doi: 10.1016/j.jht.2014.07.008. Epub 2014 Oct 6. PMID 25446519
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Jablecki CK, Andary MT, Floeter MK, Miller RG, Quartly CA, Vennix MJ, Wilson JR; American Association of Electrodiagnostic Medicine; American Academy of Neurology; American Academy of Physical Medicine and Rehabilitation. Practice parameter: Electrodiagnostic studies in carpal tunnel syndrome [RETIRED]. Report of the American Association of Electrodiagnostic Medicine, American Academy of Neurology, and the American Academy of Physical Medicine and Rehabilitation. Neurology. 2002 Jun 11;58(11):1589-92. doi: 10.1212/wnl.58.11.1589. No abstract available. PMID 12058083
- [Background] Weng C, Dong H, Chu H, Lu Z. Clinical and electrophysiological evaluation of neutral wrist nocturnal splinting in patients with carpal tunnel syndrome. J Phys Ther Sci. 2016 Aug;28(8):2274-8. doi: 10.1589/jpts.28.2274. Epub 2016 Aug 31. PMID 27630413
- [Background] Oteo-Alvaro A, Marin MT, Matas JA, Vaquero J. [Spanish validation of the Boston Carpal Tunnel Questionnaire]. Med Clin (Barc). 2016 Mar 18;146(6):247-53. doi: 10.1016/j.medcli.2015.10.013. Epub 2015 Dec 10. Spanish. PMID 26683079
- [Background] Healy A, Farmer S, Pandyan A, Chockalingam N. A systematic review of randomised controlled trials assessing effectiveness of prosthetic and orthotic interventions. PLoS One. 2018 Mar 14;13(3):e0192094. doi: 10.1371/journal.pone.0192094. eCollection 2018. PMID 29538382